CLINICAL TRIAL: NCT07142096
Title: WinQ : a Window of Opportunity Study With MitoQ in Breast Cancer
Acronym: WinQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WinQ
Record Dates: First submitted 2025-07-15; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — mitoquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MitoQ supplement (Experimental)
  Interventions: Dietary Supplement: MitoQ (mitoquinol mesylate)

INTERVENTIONS:
Dietary Supplement: MitoQ (mitoquinol mesylate) — Dietary supplement course before surgery or chemo/radio-therapy

SUMMARY:
The purpose of the study is to validate biomarkers in blood and tumor biopsy in patients with Triple Negative Breast Cancer, after a course of MitoQ treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria for study entry:
* Signed Informed Consent Form (ICF)
* Ability to comply with protocol, in the investigator's judgment
* Women aged > 18 years (no limit of age)
* ECOG performance status of 0 or 1
* Histologically documented TNBC (negative ER, - PR and HER2, status); HER2 negativity will be defined using ISH or IHC assays per ASCO/CAP criteria [1] and ER/PR negativity will be defined with < 10% tumor cells with ER/PgR staining using IHC. Patients with multifocal, multicentric or bilateral tumors are eligible, provided all discrete lesions are sampled and confirmed as triple- negative.
* Histologically confirmed invasive breast carcinoma
* Patient agreement to undergo appropriate systemic and surgical management after completion of window treatment
* Adequate hematologic and end-organ function, as defined by the following laboratory results obtained within 14 days prior to the first study treatment:
* ANC > 1500 cells/µL (without granulocyte colony-stimulating factor support within
* 2 weeks prior to Cycle 1, Day 1)
* Platelet count > 100,000/µL (without transfusion within 2 weeks prior to Cycle 1, Day 1)
* Hemoglobin > 9.0 g/dL
* Patients may be transfused to meet this criterion.
* AST, ALT, and alkaline phosphatase
* < 2.5 x the upper limit of normal (ULN)
* Serum bilirubin < 1.0 x ULN
* Patients with known Gilbert disease: serum bilirubin level < 3 x ULN
* For patients not receiving therapeutic anticoagulation: INR or aPTT < 1.5 x ULN within 14 days prior to initiation of study treatment
* For patients receiving therapeutic anticoagulation: INR or aPTT within therapeutic limits for at least 1 week immediately prior to initiation of study treatment
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen and stable INR during the 14 days immediately preceding initiation of study treatment
* Creatinine clearance > 30 mL/min (calculated using the Cockcroft-Gault formula)
* Serum albumin > 2.5 g/dL
* Beta-HCG negative if applicable (cfr infra)
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or at least 20 unstained slides, with an associated pathology report documenting ER, PR, and HER2 negativity. Tumor tissue should be of good quality based on total and viable tumor content.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year, during the treatment period and for at least 1 month after the last dose of MitoQ.
* A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (> 12 continuous months of amenorrhea with no identified cause other than menopause) and has not undergone surgical sterilization (removal of ovaries and/or uterus).
* Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established, hormone-releasing intrauterine devices (IUDs), and copper IUDs.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Women who are not postmenopausal (> 12 months of non-therapy-induced amenorrhea) or have undergone a sterilization procedure must have a negative serum pregnancy test result within 14 days prior to initiation of study food supplement.

Exclusion Criteria:

* Men
* Prior systemic therapy for treatment and prevention of the current breast cancer
* Known allergy or hypersensitivity to MitoQ
* Known active viral hepatitis
* Known human immunodeficiency virus infection with detectable viral load
* Active tuberculosis
* Severe infections within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of a food supplement or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Pregnant or lactating, or intending to become pregnant during the study Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Patients included in the study should not be under fertility preservation procedures because of the unknown effect of the treatment during human pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Biomarkers expression | Throughout the entire study, approximately during 12 months
  To assess the expression of biomarkers in fresh blood and tumor tissue, after a course of MitoQ, with RNAseq and RT-qPCR techniques
Lymphocyte tumor infiltration | Throughout the entire study, approximately during 12 months
  To asses lymphocytes infiltration by immunohistochemistry
Oxidative stress | Throughout the entire study, approximately during 12 months
  To asses the expression of biomarkers linked to oxidative stress in plasma

CONTACTS AND LOCATIONS:
Overall Officials: François Duhoux, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No